CLINICAL TRIAL: NCT04130568
Title: Translation and Adaptation of Learning Organisation Survey for French Speaking Countries
Status: Completed | Type: Observational
Sponsor: Moroccan Society of Surgery (Other)
Collaborators: Institut National d'Oncologie Sidi Mohammed Ben Abdellah (Unknown)
Responsible Party: Principal Investigator, Amine Souadka, professor, Moroccan Society of Surgery
Other Study IDs: INO_Survey
Record Dates: First submitted 2019-10-14; First posted 2019-10-17 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Learning Organization

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: INO survey — Garvin's Learning organisation tool

SUMMARY:
Learning organizations need a diagnostic tool that allows them to assess how well their team, department or the entire institution is performing, that allow them identify areas of improvement. In turn, having that tool in your own language (in this case French) and adapted to your own context, gives reliability and ease of application. Health organizations are starting to use more and more tools like this that allow them to improve their learning capabilities and therefore their performance.

Aim : described the translation of Garvin's et al. Learning Organization Survey into French to evaluate french speaking health organizations.

DETAILED DESCRIPTION:
The translation and adaptation of the survey was carried out following the steps that are recommended internationally for translation, back-translation, evaluation of translations by a commission of judges, cultural adequacy by commission of experts and, finally, a pilot test of the pre-final version.

Translation and Back-translation The first step in the process was the translation of the English LO survey by Garvin et al. (En1) based on the modified Brislin reverse translation technique.

During the translation, it was necessary to adapt some terms to maintain the same meaning as the original.

During the back-translation of the survey, no items were found that needed alteration.

The translated and back translated versions of the survey we ll be presented to a commission of 10 multidisciplinary staff from the INO. As a final part of this process, the content validity of the questions will be verified for each item of the survey.

After the necessary adjustments comparing the original survey (En1) with the back translated version (En2) and the french draft (Fr1); the french final version (FFr) of the survey will be generated and assessed in terms of conceptual equivalence, clarity and language and forwarded to the general coordinator of the project who will indicate adjustments.

Adaptation The FFr of the survey will be presented to a commission of experts in a workshop for cultural adequacy. On the day of the meeting, All multidisciplinary groups together will finish discussing and validating the pre-final french survey by mutual agreement (PFV).

Pilot test The objective of the pilot study will be to establish whether the questionnaire can be satisfactorily understood and completed by people from the target population, composed of doctors, nurses, administrators, professors. The possibility of adjustments will be considered in case the participants had difficulty understanding or responding to some item of the instrument.

Data collection The survey will be conducted anonymously and voluntarily; It will be distributed to a random sample of INO staff members, from doctors, administrators, residents, professors, nurses, technicians, secretaries. And then collected by members of the research team during August 2019.

Descriptive variables of the population were added such as: age, sex, status, years of experience, years worked in the INO and service they serve.

Analysis

The data collected will be analysed using both Excel® and IBM SPSS Statistics V22.0.

Continuous variables will be presented with mean and standard deviations(SD). Categorical variables will presented with percentage.

Normality test of the variables will be calculated using Kolmogorov-Smirnov test of normality. Cronbach's alpha coefficients will be used to assess reliability and internal consistency for each dimension, each block and the entire survey.

ANOVA test will be used to compare descriptive statistics of different groups of profession and the different Blocks and Dimensions of the survey.

ELIGIBILITY:
Inclusion Criteria:

* (1) employees at the National institut of oncology
* (2) present on the days of the survey from the 1st to 31st August 2019 (
* 3) willing to answer anonymously to this survey. Workers who were absent or on vacation were excluded as well as support staff (security and cleaning due to their frequent rotation).

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: employees at the National institut of oncology
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Translation validation of Garvin's LO survey | 4 weeks
  Translation validation of Garvin's LO survey to French

CONTACTS AND LOCATIONS:
Locations (1):
- National Institut of Oncology, Surgical oncology department, Rabat, Morocco

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Garvin DA. Building a learning organization. Harv Bus Rev. 1993 Jul-Aug;71(4):78-91. PMID 10127041
- [Background] Akhnif E, Macq J, Idrissi Fakhreddine MO, Meessen B. Scoping literature review on the Learning Organisation concept as applied to the health system. Health Res Policy Syst. 2017 Mar 1;15(1):16. doi: 10.1186/s12961-017-0176-x. PMID 28249608